CLINICAL TRIAL: NCT06616623
Title: A Phase Ib Study of Vismodegib and Atezolizumab in Patients With Advanced Non-Small Cell Lung Cancer (ML43922)
Brief Title: Vismodegib and Atezolizumab for the Treatment of Recurrent or Metastatic Non-Small Cell Lung Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Pending ICF revision
Sponsor: Dwight Owen (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dwight Owen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23268; NCI-2024-07859 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Specimen Handling; Magnetic Resonance Spectroscopy; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (vismodegib, atezolizumab) (Experimental): Patients receive vismodegib PO daily on days 1-28 and atezolizumab IV on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the study. Some patients undergo tissue sample collection during screening and on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Vismodegib

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biospecimen Collection — Undergo tissue and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC 0449; GDC-0449; GDC0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of the combination of vismodegib and atezolizumab in treating patients with non-small cell lung cancer (NSCLC) that has come back after a period of improvement (recurrent) or has spread from where it first started (primary site) to other places in the body (metastatic). Vismodegib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving a combination of vismodegib and atezolizumab may be safe, tolerable and/or effective than either drug alone in treating patients with recurrent or metastatic NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of the combination of vismodegib and atezolizumab in patients with advanced NSCLC based upon the Common Terminology Criteria for Adverse Events (CTCAE) version 5 criteria.

SECONDARY OBJECTIVE:

I. To determine the efficacy of the combination of vismodegib and atezolizumab in patients with advanced NSCLC, including progression-free survival (PFS), objective response (ORR), disease control rate (DCR), and overall survival (OS) based on modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

EXPLORATORY OBJECTIVE:

I. To study the effect of vismodegib on the levels of M2-TAMs and CD8+ T cells within the tumor microenvironment (TME) as well as myeloid-derived suppressor cells (MDSCs) in peripheral blood of study patients.

OUTLINE:

Patients receive vismodegib orally (PO) daily on days 1-28 and atezolizumab intravenously (IV) on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood sample collection throughout the study. Some patients undergo tissue sample collection during screening and on study.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed recurrent or metastatic non-small cell carcinoma of the lung of any histology without curative options
* Measurable disease based on RECIST v1.1
* Patients must have received standard of care chemotherapy and/or immunotherapy. No limits to prior lines of therapy. Prior PD-1 and/or PD-L1 directed therapies are permitted
* Patients with adenocarcinoma and known actionable mutations with Food and Drug Administration (FDA) approved treatment options must have received all approved and standard of care treatment options (i.e. osimertinib for epidermal growth factor receptor (EGFR), alectinib for anaplastic lymphoma kinase (ALK), etc.). Mutational testing is not required for patients with squamous cell non-small cell lung carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) ≥ 1,500 /mcL without granulocyte colony-stimulating factor support
* Platelet count ≥ 100,000 /uL without transfusion
* Hemoglobin ≥ 90 g/L (9 g/dL) patients may be transfused to meet this criterion
* Measured or calculated creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 mL/min for subject with creatinine levels ≤ 1.5 x institutional upper limit of normal (ULN)
* Serum total bilirubin ≤ 1.5 x ULN with the following exception:

  * Patients with known Gilbert disease: serum bilirubin ≤ 3 x ULN
* Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x ULN with the following exceptions:

  * Patients with documented liver metastases: AST and ALT ≤ 5 x ULN
  * Both values must be in the specified range
* Alkaline phosphatase (ALP) ≤ 2.5 x ULN with the following exceptions:

  * Patients with documented liver or bone metastases: ALP ≤ 5 x ULN
* Albumin ≥ 2.5 g/dL
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy

  * As long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy

  * As long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Anticipated life expectancy of ≥ 3 months
* Willing to comply with study procedures
* Female subject of childbearing potential will have a serum pregnancy test at screening. Urine pregnancy tests will be performed at specified subsequent visits. If a urine pregnancy test is positive, it must be confirmed by a serum pregnancy test
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab and 24 months after the final dose of vismodegib. Women must refrain from donating eggs during this same period
  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirement
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, for 5 months from last atezolizumab dose and 24 months after the final dose of vismodegib, as defined below:

  * With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and, for 5 months from last atezolizumab dose and 24 months after the final dose of vismodegib to avoid exposing the embryo. Men must refrain from donating sperm during this same period
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of preventing drug exposure
* Be willing and able to understand and sign the written informed consent document
* Availability of a recent formalin-fixed, paraffin-embedded (FFPE) tumor tissue block. A recently obtained archival FFPE tumor tissue block (if an FFPE tissue block cannot be provided, 15 unstained slides (10 minimum) will be acceptable) from a primary or metastatic tumor resection or biopsy can be provided if it was obtained within 1 year of trial screening
* Be willing to provide tissue from an on-treatment fine needle aspiration (FNA) or core biopsy of a tumor lesion. Subjects must consent to on-treatment biopsy prior to initiation of clinical trial, however subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may still continue on study
* Negative HIV test at screening with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count > 200/uL, and have an undetectable viral load
* Negative total hepatitis B core antibody (HBcAb) test at screening. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening

  * The HCV RNA test must be performed for patients who have a positive HCV antibody test

Exclusion Criteria:

* Active autoimmune disease requiring treatment or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are stable on thyroid-replacement hormone are eligible for the study
  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover ≤ 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at doses > 10 mg prednisone or equivalent or other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment
* Cirrhosis (Child-Pugh B or worse) or cirrhosis with history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Has symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with asymptomatic CNS lesions will be eligible if considered appropriate by the treating physician. Subjects with previously treated brain metastases may participate provided they have had a stable neurological status for at least 2 weeks after completion of definitive therapy

  * Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:

    * Measurable disease, per RECIST v1.1, must be present outside the CNS
    * The patient has no history of intracranial hemorrhage or spinal cord hemorrhage
    * The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment
    * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease
    * If the patient is receiving anti-convulsant therapy, the dose is considered stable
* Pregnancy or breastfeeding or intention of becoming pregnant during study treatment or within 5 months for atezolizumab or within 24 months after the final dose of vismodegib.

  * Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Known active tuberculosis (specific testing is only needed if clinically indicated)
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
* Prior allogeneic stem cell or solid organ transplantation
* Live, attenuated vaccines (e.g., FluMist®) are prohibited within 4 weeks prior to initiation of study treatment, during treatment with atezolizumab, and for 5 months after the last dose of atezolizumab
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Any patient who experience unacceptable toxicity on prior checkpoint inhibitor therapy:

  * ≥ grade 3 adverse event (AE) related to checkpoint inhibitor
  * ≥ grade 2 immune-related AE associated with checkpoint inhibitor
  * CNS, ocular or cardiac AE of any grade related to checkpoint inhibitor

    * NOTE: Patients with a prior endocrine AE are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years
  Will be the measured using the Common Terminology Criteria for Adverse Events version 5 criteria. Frequency and severity of AEs and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Incidence of dose limiting toxicity | Up to cycle 1 (1 cycle = 28 days)
  Will be the measured using the Common Terminology Criteria for Adverse Events version 5 criteria. Frequency and severity of AEs and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.

SECONDARY OUTCOMES:
Objective response rate | Up to 2 years
  Will be calculated and exact binomial 95% confidence interval (CI) will be provided.
Disease control rate | Up to 2 years
  Will be calculated and exact binomial 95% CI will be provided.
Overall survival (OS) | From initiation of therapy to death, or censored at last follow-up date if the subject is alive, assessed up to 2 years
  Kaplan-Meier methods will be used to estimate OS with 95% CI.
Progression free survival (PFS) | From initiation of therapy to the time of Response Evaluation Criteria in Solid Tumors progression or death, assessed up to 2 years
  Kaplan-Meier methods will be used to estimate PFS with 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Dwight H Owen, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu